CLINICAL TRIAL: NCT06332170
Title: ARTEMIS-101: A Phase 1, Open-label, Multi-center Study to Evaluate Safety, Tolerability, Pharmacokinetics and Efficacy of Intravenous Administration of HS-20093 in Combination With Other Anti-cancer Agents in Patients With Advanced Solid Tumors
Brief Title: ARTEMIS-101: A Study of HS-20093 Combinations in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HS-20093-103
Record Dates: First submitted 2024-03-18; First posted 2024-03-27 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Cisplatin; Carboplatin; Cetuximab; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1a (Experimental): HS-20093 and Adebrelimab
  Interventions: Drug: HS-20093; Drug: Adebrelimab
- Cohort 1b (Experimental): HS-20093, Adebrelimab and Cisplatin/ Carboplatin
  Interventions: Drug: HS-20093; Drug: Adebrelimab; Drug: Cisplatin/ Carboplatin
- Cohort 2a (Experimental): HS-20093 and Cetuximab
  Interventions: Drug: HS-20093; Drug: Cetuximab
- Cohort 2b (Experimental): HS-20093, Cetuximab and Cisplatin/ Carboplatin
  Interventions: Drug: HS-20093; Drug: Cisplatin/ Carboplatin; Drug: Cetuximab
- Cohort 3a (Experimental): HS-20093 and Enzalutamide
  Interventions: Drug: HS-20093; Drug: Enzalutamide

INTERVENTIONS:
Drug: HS-20093 — administered as an IV infusion
Drug: Adebrelimab — administered as an IV infusion
  Arms: Cohort 1a; Cohort 1b
Drug: Cisplatin/ Carboplatin — administered as an IV infusion
  Arms: Cohort 1b; Cohort 2b
Drug: Cetuximab — administered as an IV infusion
  Arms: Cohort 2a; Cohort 2b
Drug: Enzalutamide — 160mg once daily (QD) orally
  Arms: Cohort 3a

SUMMARY:
HS-20093 is a fully humanized IgG1 antibody-drug conjugate (ADC) which specifically binds to B7-H3, a target wildly expressed on solid tumor cells. The objectives of this study are to investigate the safety, tolerability, pharmacokinetics and anti-tumor activity of HS-20093 in combination with other anti-cancer agents in patients with advanced solid tumor patients.

DETAILED DESCRIPTION:
This is a phase 1, open-label, multi-center, dose-escalation and expansion, phase 1 study in Chinses subjects with advanced solid tumors. This study is in design allowing assessment of safety, tolerability, pharmacokinetics and anti-tumor activity of HS-20093 in combination with other anti-cancer agents.

A total of 5 combination-treatments will be carried out in 3 cohorts. The target population of dose escalation part is patients have progressed on or intolerant to available standard therapies, and the dose expansion part will enroll patients who have not received prior treatment for advanced/metastatic disease.

All patients will be carefully followed for adverse events during the study treatment and for 90 days after the last dose of study drug. Subjects will be permitted to continue therapy with assessments for progression if the product is well tolerated and sustained clinical benefit exists.

ELIGIBILITY:
Inclusion Criteria:

* At least age of 18 years at screening;
* Histologically or cytologically confirmed, locally advanced or metastatic solid tumors

  1. Dose escalation part will enroll advanced solid tumor for which standard treatment has proven ineffective or unavailable or intolerable.
  2. Dose expansion part will enroll patients who have not received prior treatment for advanced/metastatic disease.
* least one extra-cranial measurable lesion according to RECIST 1
* Agree to provide fresh or archival tumor tissue
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0~1
* Life expectancy >= 12 weeks
* Agree to use medically accepted methods of contraception
* Men or women should be using adequate contraceptive measures throughout the study;
* Females subjects must not be pregnant at screening or have evidence of non-childbearing potential
* Signed and dated Informed Consent Form

Exclusion Criteria:

* Any of the following would exclude the subject from participation in the study:

treatment with any of the following: Previous or current treatment with B7-H3 targeted therapy Intolerable for any PD-L1 inhibitor, cetuximab, enzalutamide and cisplatin/ carboplatin Cytotoxic chemotherapy, investigational agents and anticancer drugs within 14 days prior to the first scheduled dose of HS-20093 Prior treatment with a monoclonal antibody within 28 days prior to the first scheduled dose of HS-20093 Radiotherapy with a limited field of radiation for palliation within 2 weeks, or patients received more than 30% of the bone marrow irradiation, or large-scale radiotherapy within 4 weeks prior to the first scheduled dose of HS-20093 Major surgery within 4 weeks prior to the first scheduled dose of HS-20093

* Subjects with previous or concurrent malignancies
* Inadequate bone marrow reserve or organ dysfunction
* Evidence of cardiovascular risk
* Evidence of current severe or uncontrolled systemic diseases
* Evidence of mucosal or internal bleeding within 1 month prior to the first scheduled dose of HS-20093
* Known active infection requiring antibodies treatment within 2 weeks, or severe infection within 4 weeks prior to the first scheduled dose of HS-20093
* Subjects with current infectious diseases
* History of neuropathy or mental disorders
* Pregnant or lactating female
* History of severe hypersensitivity reaction, severe infusion reaction or idiosyncrasy to drugs chemically related to HS-20093 or any of the components of HS-20093
* Unlikely to comply with study procedures, restrictions, and requirements in the opinion of the investigator
* Any disease or condition that, in the opinion of the investigator, would compromise subject safety or interfere with study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) for combination-treatments | Up to day 21 from the first dose
  To determine the MTD for further evaluation of HS-20093 with other anti-cancer agents in subjects with advanced solid tumors

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) | From the first dose through 90 days post end of treatment
  AE assessed by investigator exclusively related to subject's underlying disease or medical condition [graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0]. Any untoward medical occurrence in a clinical study participant, whether or not considered related to the medicinal product. Incidence and severity of AEs are assessed according to vital signs, laboratory variables, physical examination, electrocardiogram, etc.
Objective response rate (ORR) determined by investigators | From the first dose up to PD or withdrawal from study, whichever came first, assessed up to 24 months
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline. ORR is evaluated by the number of participants with best overall response of CR and PR (Confirmed CR/PR assessment require at least 1 repeat). For prostate cancer patients, ORR is determined by investigators according to RECIST 1.1 and Prostate Cancer Working Group 3 (PCWG3).
Disease control rate (DCR) determined by investigators | From the first dose up to PD or withdrawal from study, whichever came first, assessed up to 24 months
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline. DCR was evaluated by the number of participants with best overall response of CR, PR and stable disease (SD) [Confirmed CR/PR assessment require at least one repeat (≥4 weeks); SD shall be assessed at least 5 weeks after the first dose]. For prostate cancer patients, DCR is determined by investigators according to RECIST 1.1 and Prostate Cancer Working Group 3 (PCWG3).
Duration of response (DoR) determined by investigators | From the first dose up to PD or death, whichever came first, assessed up to 24 months
  DoR was defined as the period from the first occurrence of CR or PR to PD or death from any cause. If no PD or death after CR/PR, the cut-off date of progression-free survival (PFS) would be used [Confirmed CR/PR assessment require at least one repeat (≥4 weeks)]. For prostate cancer patients, DoR is determined by investigators according to RECIST 1.1 and Prostate Cancer Working Group 3 (PCWG3).
Progression-free survival (PFS) determined by investigators according to RECIST 1.1 | From the first dose up to PD or death, whichever came first, assessed up to 24 months
  PFS was defined as the time from random assignment or first dose to PD or death from any cause.
Overall survival (OS) | From the first dose up to death, whichever came first, assessed up to 24 months
  OS was defined as the time from random assignment or first dose to death from any cause.
Radiographic progression-free survival (rPFS) determined by investigators according to RECIST 1.1 and PCWG3 | From the first dose up to PD or death from study, whichever came first, assessed up to 24 months
  For prostate cancer patients, the rPFS is defined as the time from random assignment or first dose to the date of first documented PD per PCWG3 or death from any cause, whichever occurs first.
Time to PSA progression (TTPP) | From the first dose up to PD or withdrawal from study, whichever came first, assessed up to 24 months
  In participants with a decrease in PSA from baseline: ≥ 25% increase and an absolute increase of ≥ 2 ng/mL above the nadir value, which is confirmed by a consecutive second value obtained ≥ 3 weeks later. In participants with no decrease in PSA from baseline: ≥ 25% increase and an absolute increase of ≥ 2 ng/mL above the baseline value after 12 weeks.
Prostate-specific cancer antigen (PSA) response rate | From the first dose up to PD or withdrawal from study, whichever came first, assessed up to 24 months
  PSA response is defined as a ≥ 50% decline in PSA from baseline with PSA confirmation ≥ 3 weeks after the first documented reduction in PSA of ≥ 50%.
Time to first subsequent therapy (TFST) | From the first dose up to the imitation of subsequent therapy or death, whichever came first, assessed up to 24 months
  TFST was defined as the time from random assignment or first dose to the imitation of subsequent therapy or death.
Observed maximum plasma concentration (Cmax) of HS-20093advanced solid tumor | From pre-dose to study completion, assessed up to 24 months
  Cmax will be obtained after administration of the first dose of HS-20093
Time to reach maximum plasma concentration (Tmax) of HS-20093 | From pre-dose to study completion, assessed up to 24 months
  Tmax will be obtained after administration of the first dose of HS-20093
Terminal half-life (T1/2) of HS-20093 following the first dose | From pre-dose to study completion, assessed up to 24 months
  T1/2 will be obtained after administration of the first dose of HS-20093
Area under plasma concentration versus time curve from zero to last sampling time (AUC0-t) following the first dose of HS-20093 | From pre-dose to study completion, assessed up to 24 months
  Area under the plasma concentration versus time curve from time zero to the last sampling time when the concentration was no less than the lower limit of quantification (LLQ). AUC0-t was calculated according to the mixed log-linear trapezoidal rule.
Percentage of participants with antibodies to HS-20093 in serum | From pre-dose to study completion, assessed up to 24 months
  Serum samples were collected for the determination of anti-drug antibody (ADA) at designated time points.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided